CLINICAL TRIAL: NCT03560817
Title: Survey of Health Preferences in Cancer Patients: a Study Protocol for a Prospective, Longitudinal Cohort Using Online Survey
Brief Title: Survey of Health Preferences in Cancer Patients (QALY-Cancer)
Acronym: QALY-Cancer
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Thomas G. Poder, Principal Investigator, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Other Study IDs: 2017-1490
Record Dates: First submitted 2018-04-27; First posted 2018-06-18 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: QALY; Cost-utility analysis; Time-trade-off method; Discrete choice experiment method
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast cancer: No intervention is added with the study. Patients follow their standard treatment and respond to an online questionnaire about their health preferences.
- colorectal cancer: No intervention is added with the study. Patients follow their standard treatment and respond to an online questionnaire about their health preferences.

SUMMARY:
This study will evaluate health utilities in patients with breast or colorectal cancer.

DETAILED DESCRIPTION:
The cost-utility analysis (CUA) is an increasingly used method to help health decision-maker. The CUA uses the Quality Adjusted Life Years (QALY) that combines the length of life with the health related quality of life (HRQoL) into a single score.

In Quebec, no QALY calculation tool has been adapted to its linguistic and socio-cultural context, neither for its general population nor for a particular subpopulation, like patients with cancer.

The objectives will be to analyze the extent of the divergence in terms of health states utilities between the general population and patients with breast or colorectal cancer; to develop a QALY preference weights dataset for patients with cancer; to perform "mapping" with different health-related quality of life questionnaires by correlating SF6Dv2 with EQ-5D-5L, EORTC QLQ-C30 and FACT- G. The data will be collected with a self-administered online survey. Patients outcomes will be measured at the beginning of the chemotherapy treatment cycle and about 8 days after the start of chemotherapy. Health utilities will be measured with a hybrid method using the time-trade-off (TTO) and the discrete experimental choice (DCE) method using SF6Dv2 questionnaire for health states.

ELIGIBILITY:
Inclusion Criteria:

* to be 18 years of age or older;
* to reside in Quebec;
* have already had a chemotherapy treatment cycle;
* be on the eve of a new round of chemotherapy treatment;
* have breast or colorectal cancer

Exclusion Criteria:

* being over 80 years of age;
* not be able to complete a computer questionnaire;
* can not read or write in French;
* not be able to sign a consent form;
* the only treatment offered is surgery;
* presence of metastases to the brain;
* patient with delirium, psychosis or severe depression (i.e. chronic condition with treatment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of the Quebec population aged 18 and over who have breast cancer or colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Health utilities for SF-6Dv2 before chemotherapy | Within two days before the start of a chemotherapy treatment cycle (standard treatment; each cycle is 21 days)
  Health utilities measured by SF-6Dv2 health states using a hybrid method combining time-trade-off (TTO) and discrete choice experiment (DCE)
Health utilities for SF-6Dv2 after the start of the chemotherapy | 8 days after the start of the chemotherapy
  Health utilities measured by SF-6Dv2 health states using a hybrid method combining time-trade-off (TTO) and discrete choice experiment (DCE)

SECONDARY OUTCOMES:
Health utilities with the EuroQol five-dimensional questionnaire with five response levels (EQ-5D-5L) before chemotherapy | Within two days before the start of a chemotherapy treatment cycle (standard treatment; each cycle is 21 days)
  The EQ-5D-5L included five health dimensions with five response levels of 1 to 5. A score is calculated using an already pre-established regression equation using time-trade-off method. The health utilities range from -0.148 for the worst EQ-5D-5L state to 0.949 for the best EQ-5D-5L state.
Health related quality of life (HRQoL) scores from EORTC QLQ-C30 questionnaire before chemotherapy before chemotherapy | Within two days before the start of a chemotherapy treatment cycle (standard treatment; each cycle is 21 days)
  The EORTC QLQ-C30 questionnaire were developed by the European Organisation for Research and Treatment of Cancer (EORTC). Including 30items, evaluating five functions, nine symptoms, and the overall health status of patients with cancer. Scales will be calculated by averaging the items. Items and scales will be linearly transformed to a range of 0 to 100. A higher score indicate a better quality of life or higher symptoms.
Health related quality of life (HRQoL) scores from the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaires before chemotherapy | Within two days before the start of a chemotherapy treatment cycle (standard treatment; each cycle is 21 days)
  The survey assesses the impacts of cancer therapy in four domains: physical, social/family, emotional, and functional. It include 27 questions, each of which is answered using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Higher numbers indicate a better health state. The score will be calculated with the sum of items and score will be normalised on a scale from 0-100.
Health utilities with the EuroQol five-dimensional questionnaire with five response levels (EQ-5D-5L) after chemotherapy | 8 days after the start of the chemotherapy
  The EQ-5D-5L included five health dimensions with five response levels of 1 to 5. A score is calculated using an already pre-established regression equation using time-trade-off method. The health utilities range from -0.148 for the worst EQ-5D-5L state to 0.949 for the best EQ-5D-5L state.
Health related quality of life (HRQoL) scores from EORTC QLQ-C30 questionnaire before after chemotherapy | 8 days after the start of the chemotherapy
  The EORTC QLQ-C30 questionnaire were developed by the European Organisation for Research and Treatment of Cancer (EORTC). Including 30items, evaluating five functions, nine symptoms, and the overall health status of patients with cancer. Scales will be calculated by averaging the items. Items and scales will be linearly transformed to a range of 0 to 100. A higher score indicate a better quality of life or higher symptoms.
Health related quality of life (HRQoL) scores from the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaires after chemotherapy | 8 days after the start of the chemotherapy
  The survey assesses the impacts of cancer therapy in four domains: physical, social/family, emotional, and functional. It include 27 questions, each of which is answered using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Higher numbers indicate a better health state. The score will be calculated with the sum of items and score will be normalised on a scale from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Poder, PhD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre de recherche du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No